CLINICAL TRIAL: NCT04230577
Title: Transcranial Photobiomodulation to Improve Cognition in TBI, With Pre-/Post- fMRI Scans: A Pilot, Sham-Controlled Study
Brief Title: Photobiomodulation to Improve Cognition in TBI, With fMRI
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: VA Boston Healthcare System (U.S. Federal Agency); Vielight Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0216aVielight; 3223 (Other: VABHS)
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Traumatic Brain Injury; Closed Head Injury; Cognitive Dysfunction
Keywords: mild-moderate traumatic brain injury; TBI; Cognition; Executive Function; Attention; Memory; Photobiomodulation (PBM); Low-level Laser Therapy (LLLT); Light-Emitting Diodes (LEDs); Magnetic Resonance Imaging (MRI); functional MRI (fMRI); resting-state functional connectivity MRI (rs-fcMRI); Magnetic Resonance Spectroscopy (MRS); Post Traumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Brain Injuries, Traumatic; Head Injuries, Closed; Cognitive Dysfunction; Stress Disorders, Post-Traumatic | interventions — Therapeutics; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This study is a blinded, randomized, sham-controlled, partial-crossover study with 2 groups (n=10 per group (Sham, Real); ages 18-65). Participants are randomized by computer into group 1 or 2, in blocks of 10. At-home LED intervention is self-administered 3 times per week (20 minutes), for two 5-week series, with a one month break between series. All participants receive a Real Series of treatment at some point during the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After consent/screening participant is randomized by computer into Group 1 or Group 2 in blocks of 10. The participant, investigator and outcome assessor is blinded to Group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real LED Intervention (Active Comparator): Participants receive 15 Real (active) LED treatments with the Vielight Neuro Alpha head frame device (with intranasal). Parameters: NIR, 810nm, pulsed at 10 Hz, 50% duty cycle, synchronized for a 20-minute treatment time. Total Energy Dose per head set plus intranasal: 225 J/cm2+ 15 J/cm2 = 240 J/cm2 per 20 min LED treatment. Total Energy Dose delivered (3x/Week, 5 Weeks) = 3600 J/cm2. The light from these LEDs is not visible to the eye. There is no potential for eye damage because the LEDs are not laser light. The head frame device falls within the FDA category General Wellness, low-risk devices, and no medical claims are made. It is approved for use by the VA Boston Healthcare System Safety Committee and Institutional Review Board.
  Interventions: Device: Real LED Intervention
- Sham LED Intervention (Sham Comparator): Participants receive a series of 15 Sham (control) LED treatments with the Vielight Neuro Alpha head frame device (with intranasal) containing Sham LEDs, synchronized for a 20-minute treatment time (3x/Week, 5 Weeks). Sham and Real devices are identical in look and feel, except no photons are emitted from the Sham devices.
  Interventions: Device: Real LED Intervention; Device: Sham LED Intervention

INTERVENTIONS:
Device: Real LED Intervention — A series of Real at-home, transcranial LED treatments (3xWeek, 5 weeks), 20-minute treatment, 810nm (NIR), Vielight Neuro Alpha Head Frame Device (with NIR intranasal).
  Other Names: Light-Emitting Diode (LED) Therapy; Photobiomodulation (PBM); Vielight Neuro Alpha
Device: Sham LED Intervention — A series of Sham at-home, transcranial LED treatments (3xWeek, 5 weeks), 20-minute treatment, Vielight Neuro Alpha Head Frame Device (with intranasal) with Sham LEDs that emit no photons. Sham and Real Devices look and feel identical.
  Other Names: Control
  Arms: Sham LED Intervention

SUMMARY:
The purpose of this small, research study is to examine effectiveness of an at-home application of an experimental intervention, on thinking and memory in mild-moderate, closed-head, traumatic brain injury cases. The experimental intervention is light-emitting diode (LED) therapy, which is applied to the scalp and through the nose using a head frame device. Participants are expected to complete two, 5-week series of LED treatments, at home, 3 times a week. There will be a 1-month period between the two series. Each home treatment is 20 minutes. Participants will be trained to use the head frame device, in-office. The head frame device falls within the FDA category General Wellness, low-risk devices, and no medical claims are made. A two-hour paper and pencil testing (4 visits) and a one-hour MRI (3 visits) will be administered before and after each treatment series. Participants may be in the study for about 4 months. This study is supported by Vielight, Inc., Hayward, CA/ Toronto, Canada

DETAILED DESCRIPTION:
Objectives: This small study examines effectiveness of an at-home experimental intervention that utilizes near-infrared (NIR) wavelengths of light (810nm) applied to the scalp, using light-emitting diodes (LEDs), to improve brain function. LEDs may directly improve the cellular activity of brain tissue that has been damaged by brain trauma. The intervention involves two series of 15 treatments, which are self-administered, at-home. Neuropsychological testing and structural and functional MRI (fMRI) scans will be administered to examine behavioral and brain changes before and after a series of LED treatments. MRI scans will examine some mechanism of LED intervention including changes in blood flow, functional connectivity and neurochemicals.

Research Design: This study is a blinded, randomized, sham-controlled, partial-crossover study, with 2 groups (n=10 per group (Sham, Real); ages 18-65). Participants are randomized, by computer into groups. At-home LED intervention is self-administered 3 times per week (20 minutes), for two 5-week series, with a one-month break between series. Group 1 receives both a series of Sham and a series of Real treatments and Group 2 receives two series of Real treatments. All participants will receive at least one series of Real treatments during participation.

Methods and General Study Procedure: Twenty veterans with traumatic brain injury, 18-65 years old, who are at least 6-months post- the latest mild-moderate traumatic brain injury (TBI) will be studied. A 1-hour, In-office neuropsychological (NP) screening, after consenting, will determine study eligibility and ensure participants meet the inclusion/exclusion criteria. Participants may be in the study for about 4 months.

Device Parameters: Vielight Neuro Alpha head frame device, NIR, 810nm, pulsed at 10 Hz, 50% duty cycle, 20-minute treatment with automatic shutoff. Total Energy Dose per head set plus intranasal: 225 J/cm2+ 15 J/cm2 = 240 J/cm2 per 20 min LED treatment. Total Energy Dose delivered (3x/Week, 5 Weeks) = 3600 J/cm2. The light from these LEDs is not visible to the eye. There is no potential for eye damage because the LEDs are not laser light.

Sham and Real devices are identical in look and feel, except no photons are emitted from the Sham devices. The head frame device falls within the FDA category General Wellness, low-risk devices, and no medical claims are made. It is approved for use by the VA Boston Healthcare System Safety and Human Subjects Committees.

Training: Each participant is assigned his/her own LED head frame device for hygiene reasons. The assigned device will be provided to each participant at a 1-hour in-office training session, after the first Neuropsychological (NP) Testing. Training that includes both verbal and written instructions will be provided, along with demonstration of use of the device. A treatment log, storage box and alcohol wipes for cleaning are provided. The first treatment is completed at the training session.

For each series of LED treatments, a 20-minute, LED treatment is completed at home, 3 times per week (Monday, Wednesday, and Friday), for 5 weeks. There must be at least 48 hours between treatments. There will be a total of 15 treatments in each series. The specific time of day is at the participant's convenience. Missed treatments will be completed at the end of the 5-week series, so all participants will complete all 15 LED treatments. If more than 1 treatment session in a week is not completed, due to unforeseen circumstances, the participant may be withdrawn from the study.

A staff person will telephone each participant weekly, to fill out a questionnaire about the intervention including inquiring if the LED treatments are being performed, if the treatment log sheets are being filled out, and note if there are any questions, concerns or problems.

Neuropsychological Testing: All NP testing is completed at the VA Boston Healthcare System, Jamaica Plain Campus, Boston, MA.

NP tests are administered at four time points (pre- intervention, with follow-up testing at 1 week and 1 month post- series 1, and 1 week post- series 2): The California Verbal Learning Test (CVLT), Long-Delay Free Recall (LDFR) is the Primary Outcome Measure which examines verbal learning, organization and memory. The subtest LDFR, CVLT-II specifically assesses long-delay (20 min), verbal memory, which can be affected after mild-moderate brain injury. Other NP, Psychosocial and General Health measures are considered Secondary Outcome Measures. To avoid practice effects, alternate versions of the NP tests will be used at the Post- LED testing times, when feasible.

Imaging will be conducted on the 3T Philips MRI system located at the Boston University Center for Biomedical Imaging (BU CBI). One-hour scans are acquired at 3 time points, in all participants. No contrast or x-rays are used.

Participants are permitted to have an MRI brain scan, if it has been determined at Entry, that MRI scanning would be safe using an MRI safety checklist. On the day of the MRI scan at the BU CBI, the BU Safety Checklist will also be reviewed before any scanning will occur. The light therapy portion of the study may be completed, even if participants cannot undergo MRI scanning for medical or safety reasons.

Functional MRI: resting-state functional-connectivity Magnetic Resonance Imaging (rs-fc MRI) is the Primary Imaging Outcome Measure. Rs-fc MRI examines the correlation of low frequency signal between voxels in the brain in different areas. Rs-fc MRI abnormalities have been shown in mild-moderate TBI cases. Other imaging sequences are considered exploratory measures. These will provide information on brain structure, blood flow and neurochemicals.

Statistical Analysis Plan

Neuropsychological, Psychosocial, and Health Data Analysis: VA Biostatistician, Robert Lew, PhD.

This study has two 5-week Series (I and II). In Series I, 10 subjects will be assigned to (A), and 10 assigned to (B). In Series II, all remaining A-subjects will continue on A, and all remaining B subjects will switch to A. Switching increases power and reduces dropout. For subjects in treatment B and then A, the model will include a compound symmetry correlation term (r=0.30). Treated subjects are Series I A; and Series II, switch-to-A.

To test if the change between consecutive times, delta, is positive for A, we will model the response, as measured by the CVLT, LDFR in mixed design random effects model of analysis. The formal hypothesis test is a linear contrast, a t-test that assumes an effect size of 0.5. For all Secondary Outcome Measures, exploratory analyses will confirm or not the results for primary hypothesis, CVLT, LDFR. A mixed design random effects model should enable handling of missing data points.

Statistical Analyses for MRI/fMRI data MRI data will be analyzed using Matlab, parametric statistics, and available standard Imaging software. All analyses will be parametric and corrections for multiple comparisons will be made.

Between group comparison of MRI data for the active vs. control groups (at time points T1-T3) will be completed.

Longitudinal impact of treatment over time on MRI scans Analyses will be a within-subject design, which compares changes pre- to 1-week post- and 1-month post- Series 1 intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Must have had one (or more) closed-head, traumatic brain injuries
* Loss of consciousness 24 hours or less; or no loss of consciousness/ A period of altered mental status (post-traumatic amnesia)/mental confusion for 24 hours or less
* Must be able to come to VA Boston Healthcare System, Jamaica Plain Campus for testing visits and Boston University Center for Biomedical Imaging, Boston University School of Medicine for MRI scans

Must meet the following Screening requirements:

* Participants must score at least 2 SD below normal on at least 1 of the NP tests; or 1 SD below on at least 2 of these NP tests administer at Entry testing: Trail Making Test A & B; Controlled Oral Word Association Test (COWAT/FAS); California Verbal Learning Test II; DKEFS Color-Word Interference Test (Stroop).

Exclusion Criteria:

* Diagnosis of a neurological disease such amyotrophic lateral sclerosis (ALS), Parkinson's, Alzheimer's disease
* History of craniotomy or craniectomy
* A current life-threatening disease such as cancer
* Disease requiring organ transplant
* A severe mental disorder such as schizophrenia, bipolar disorder (not associated with clinically diagnosed PTSD)
* Current substance abuse or active treatment; within the last 6 months
* The Test of Memory Malingering is administered at screening; Participants must not have scores that indicate evidence of malingering, a score of less than 45 on either Part 1 or 2 would show evidence of malingering, with the following exception: If a participant fails Trial 1, but does not fail Trial 2, he/she would not be excluded if he/she also show evidence of poor learning on other NP Screening tests, such as the CVLT. If he/she fails Trial 2, alone, or Trial 1 and Trial 2, then this would exclude the participant from the study.
* Self-reported pain questionnaires (VAS Pain Rating and the Short Form McGill Pain Questionnaire) are also administered. Participants may not have a level of pain greater than 7/10 on VAS or 38/50 on the McGill pain questionnaires at the time of screening.

Exclusion for Magnetic Resonance Imaging Only

* A BU MRI safety screening form will be reviewed at the time of study screening, as well as at each MRI scan appointment to ensure the participant can safely have an MRI. Participants must tell the investigator about any operations and any metal in his/her body, so it can be decided if it is safe for you to proceed with the scan.

Participants cannot have a MRI scan:

* if pregnant.
* if he/she has pacemakers, ear implants, shrapnel injuries, or other types of metal or electric device in their body

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-07 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
CVLT-II, Long Delay Free Recall 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  California Verbal Learning Test-II Long Delay (20 mins) Free Recall; Measures Verbal Memory Min score of 0 and a max score of 16; higher score = better outcome. After a 20 minute delay (other tasks run during this delay), participant is asked to recall items from List A. Total is number of words recalled.
  Alternate lists are used at each testing timepoint to avoid practice effect
CVLT-II, Long Delay Free Recall 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  California Verbal Learning Test-II Long Delay (20 mins) Free Recall; Measures Verbal Memory Min score of 0 and a max score of 16; higher score = better outcome. After a 20 minute delay (other tasks run during this delay), participant is asked to recall items from List A. Total is number of words recalled.
  Alternate lists are used at each testing timepoint to avoid practice effect
CVLT-II, Long Delay Free Recall 3 | Change from 1-Week to 1-Month after Series 1
  California Verbal Learning Test-II Long Delay (20 mins) Free Recall; Measures Verbal Memory Min score of 0 and a max score of 16; higher score = better outcome. After a 20 minute delay (other tasks run during this delay), participant is asked to recall items from List A. Total is number of words recalled.
  Alternate lists are used at each testing timepoint to avoid practice effect
CVLT-II, Long Delay Free Recall 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  California Verbal Learning Test-II Long Delay (20 mins) Free Recall; Measures Verbal Memory Min score of 0 and a max score of 16; higher score = better outcome. After a 20 minute delay (other tasks run during this delay), participant is asked to recall items from List A. Total is number of words recalled.
  Alternate lists are used at each testing timepoint to avoid practice effect

SECONDARY OUTCOMES:
CVLT-II, Short Delay Free Recall 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  California Verbal Learning Test-II Immediate Free Recall; Measures Verbal Memory Min score of 0 and a max score of 16; higher score = better outcome Participant is asked to recall items from List A. Total is number of words recalled.
CVLT-II, Short Delay Free Recall 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  California Verbal Learning Test-II Immediate Free Recall; Measures Verbal Memory Min score of 0 and a max score of 16; higher score = better outcome Participant is asked to recall items from List A. Total is number of words recalled.
CVLT-II, Short Delay Free Recall 3 | Change from 1-Week to 1-Month after Series 1
  California Verbal Learning Test-II Immediate Free Recall; Measures Verbal Memory Min score of 0 and a max score of 16; higher score = better outcome Participant is asked to recall items from List A. Total is number of words recalled.
CVLT-II, Short Delay Free Recall 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  California Verbal Learning Test-II Immediate Free Recall; Measures Verbal Memory Min score of 0 and a max score of 16; higher score = better outcome Participant is asked to recall items from List A. Total is number of words recalled.
CVLT-II, Short Delay Cued Recall 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  California Verbal Learning Test-II Immediate Cued Recall; Measures Verbal Memory Participants are asked to immediately recall items from a list, but are given cues by category. (4 categories, 4 items each). Total is score across all 4 categories.
CVLT-II, Short Delay Cued Recall 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  California Verbal Learning Test-II Immediate Cued Recall; Measures Verbal Memory Participants are asked to immediately recall items from a list, but are given cues by category. (4 categories, 4 items each). Total is score across all 4 categories.
CVLT-II, Short Delay Cued Recall 3 | Change from 1-Week to 1-Month after Series 1
  California Verbal Learning Test-II Immediate Cued Recall; Measures Verbal Memory Participants are asked to immediately recall items from a list, but are given cues by category. (4 categories, 4 items each). Total is score across all 4 categories.
CVLT-II, Short Delay Cued Recall 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  California Verbal Learning Test-II Immediate Cued Recall; Measures Verbal Memory Participants are asked to immediately recall items from a list, but are given cues by category. (4 categories, 4 items each). Total is score across all 4 categories.
CVLT-II, Long Delay Cued Recall 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  California Verbal Learning Test-II Long Delay (20 minutes) Cued Recall; Measures Verbal Memory Participants are asked to immediately recall items from a list, but are given cues by category. (4 categories, 4 items each). Total is score across all 4 categories.
CVLT-II, Long Delay Cued Recall 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  California Verbal Learning Test-II Long Delay (20 minutes) Cued Recall; Measures Verbal Memory Participants are asked to immediately recall items from a list, but are given cues by category. (4 categories, 4 items each). Total is score across all 4 categories.
CVLT-II, Long Delay Cued Recall 3 | Change from 1-Week to 1-Month after Series 1
  California Verbal Learning Test-II Long Delay (20 minutes) Cued Recall; Measures Verbal Memory Participants are asked to immediately recall items from a list, but are given cues by category. (4 categories, 4 items each). Total is score across all 4 categories.
CVLT-II, Long Delay Cued Recall 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  California Verbal Learning Test-II Long Delay (20 minutes) Cued Recall; Measures Verbal Memory Participants are asked to immediately recall items from a list, but are given cues by category. (4 categories, 4 items each). Total is score across all 4 categories.
CVLT-II, Total Trials 1-5 _1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  California Verbal Learning Test-II, Total Trials 1-5; Measures Learning/Memory over 5 consecutive trials; with a min score of 0 and a max score of 80; higher score = better outcome Participant must immediately recall words from a 16 word list read aloud by the examiner. The same list is presented for each of the 5 trials. Total across 5 trials is scored.
CVLT-II, Total Trials 1-5 _2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  California Verbal Learning Test-II, Total Trials 1-5; Measures Learning/Memory over 5 consecutive trials; with a min score of 0 and a max score of 80; higher score = better outcome Participant must immediately recall words from a 16 word list read aloud by the examiner. The same list is presented for each of the 5 trials. Total across 5 trials is scored.
CVLT-II, Total Trials 1-5 _3 | Change from 1-Week to 1-Month after Series 1
  California Verbal Learning Test-II, Total Trials 1-5; Measures Learning/Memory over 5 consecutive trials; with a min score of 0 and a max score of 80; higher score = better outcome Participant must immediately recall words from a 16 word list read aloud by the examiner. The same list is presented for each of the 5 trials. Total across 5 trials is scored.
CVLT-II, Total Trials 1-5 _4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  California Verbal Learning Test-II, Total Trials 1-5; Measures Learning/Memory over 5 consecutive trials; with a min score of 0 and a max score of 80; higher score = better outcome Participant must immediately recall words from a 16 word list read aloud by the examiner. The same list is presented for each of the 5 trials. Total across 5 trials is scored.
Color-Word Interference (Stroop) Test, Trial 3 _1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Delis-Kaplan Executive Function (DKEFS), Color-Word Interference Test; also known as the Stroop test; Trial 3 is a measure of Inhibition.
  Measures Attention/Executive Function; inhibition Measure is Reaction Time lower = better outcome Trial 3 (Inhibition): Name the color ink each word is printed in for a series of words, as quickly as possible.
Color-Word Interference (Stroop) Test, Trial 3 _2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Delis-Kaplan Executive Function (DKEFS), Color-Word Interference Test; also known as the Stroop test; Trial 3 is a measure of Inhibition.
  Measures Attention/Executive Function; inhibition Measure is Reaction Time lower = better outcome Trial 3 (Inhibition): Name the color ink each word is printed in for a series of words, as quickly as possible.
Color-Word Interference (Stroop) Test, Trial 3 _3 | Change from 1-Week to 1-Month after Series 1
  Delis-Kaplan Executive Function (DKEFS), Color-Word Interference Test; also known as the Stroop test; Trial 3 is a measure of Inhibition.
  Measures Attention/Executive Function; inhibition Measure is Reaction Time lower = better outcome Trial 3 (Inhibition): Name the color ink each word is printed in for a series of words, as quickly as possible.
Color-Word Interference (Stroop) Test, Trial 3 _4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Delis-Kaplan Executive Function (DKEFS), Color-Word Interference Test; also known as the Stroop test; Trial 3 is a measure of Inhibition.
  Measures Attention/Executive Function; inhibition Measure is Reaction Time lower = better outcome Trial 3 (Inhibition): Name the color ink each word is printed in for a series of words, as quickly as possible.
Color-Word Interference (Stroop) Test, Trial 4 _1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Delis-Kaplan Executive Function (DKEFS), Color-Word Interference Test; also known as the Stroop test; Trial 4 is a measure of executive function: Inhibition/switching.
  Measures Attention/Executive Function; inhibition/switching Measure is Reaction Time lower = better outcome Trial 4 (Inhibition and Switching): Name the color of the ink, however if there is a box around the word, read the word, as quickly as possible
Color-Word Interference (Stroop) Test, Trial 4 _2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Delis-Kaplan Executive Function (DKEFS), Color-Word Interference Test; also known as the Stroop test; Trial 4 is a measure of executive function: Inhibition/switching.
  Measures Attention/Executive Function; inhibition/switching Measure is Reaction Time lower = better outcome Trial 4 (Inhibition and Switching): Name the color of the ink, however if there is a box around the word, read the word, as quickly as possible
Color-Word Interference (Stroop) Test, Trial 4 _3 | Change from 1-Week to 1-Month after Series 1
  Delis-Kaplan Executive Function (DKEFS), Color-Word Interference Test; also known as the Stroop test; Trial 4 is a measure of executive function: Inhibition/switching.
  Measures Attention/Executive Function; inhibition/switching Measure is Reaction Time lower = better outcome Trial 4 (Inhibition and Switching): Name the color of the ink, however if there is a box around the word, read the word, as quickly as possible
Color-Word Interference (Stroop) Test, Trial 4 _4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Delis-Kaplan Executive Function (DKEFS), Color-Word Interference Test; also known as the Stroop test; Trial 4 is a measure of executive function: Inhibition/switching.
  Measures Attention/Executive Function; inhibition/switching Measure is Reaction Time lower = better outcome Trial 4 (Inhibition and Switching): Name the color of the ink, however if there is a box around the word, read the word, as quickly as possible
Delis-Kaplan Executive Function Trails (Condition 2) 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Number Sequencing; measures Attention/Executive Function, Sequencing, Visual Scanning Measure is Reaction Time with lower = better outcome Connect the numbers in consecutive order from 1 to 16, as quickly as possible.
Delis-Kaplan Executive Function Trails (Condition 2) 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Number Sequencing; measures Attention/Executive Function, Sequencing, Visual Scanning Measure is Reaction Time with lower = better outcome Connect the numbers in consecutive order from 1 to 16, as quickly as possible.
Delis-Kaplan Executive Function Trails (Condition 2) 3 | Change from 1-Week to 1-Month after Series 1
  Number Sequencing; measures Attention/Executive Function, Sequencing, Visual Scanning Measure is Reaction Time with lower = better outcome Connect the numbers in consecutive order from 1 to 16, as quickly as possible.
Delis-Kaplan Executive Function Trails (Condition 2) 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Number Sequencing; measures Attention/Executive Function, Sequencing, Visual Scanning Measure is Reaction Time with lower = better outcome Connect the numbers in consecutive order from 1 to 16, as quickly as possible.
Delis-Kaplan Executive Function Trails (Condition 4) 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Number and Letter Sequencing; measures Attention/Executive Function, Sequencing, Visual Scanning Measure is Reaction Time with lower = better outcome Alternate connecting numbers and letters in consecutive order from 1 to P (1-A-2-B…) as quickly as possible.
Delis-Kaplan Executive Function Trails (Condition 4) 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Number and Letter Sequencing; measures Attention/Executive Function, Sequencing, Visual Scanning Measure is Reaction Time with lower = better outcome Alternate connecting numbers and letters in consecutive order from 1 to P (1-A-2-B…) as quickly as possible.
Delis-Kaplan Executive Function Trails (Condition 4) 3 | Change from 1-Week to 1-Month after Series 1
  Number and Letter Sequencing; measures Attention/Executive Function, Sequencing, Visual Scanning Measure is Reaction Time with lower = better outcome Alternate connecting numbers and letters in consecutive order from 1 to P (1-A-2-B…) as quickly as possible.
Delis-Kaplan Executive Function Trails (Condition 4) 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Number and Letter Sequencing; measures Attention/Executive Function, Sequencing, Visual Scanning Measure is Reaction Time with lower = better outcome Alternate connecting numbers and letters in consecutive order from 1 to P (1-A-2-B…) as quickly as possible.
Benton Visual Memory Test; Trial 1 Immediate Recall 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Immediate Recall for Visuospatial memory Min 0 and max 36; higher score better outcome Participant is presented with 6 figures. They are given 10 secs to view 6 pictures. Immediately asked to recall and draw the figures.
  Up to 2 points per figure. Scoring based on accuracy and placement of figure parts: A score of 0, 1 recognizable and incorrectly placed, 1 accurate or correctly placed or 2 both accurate and correctly placed; 0 is given if part is omitted or unrecognizable.
  Total possible 12 points
Benton Visual Memory Test; Trial 1 Immediate Recall 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Immediate Recall for Visuospatial memory Min 0 and max 36; higher score better outcome Participant is presented with 6 figures. They are given 10 secs to view 6 pictures. Immediately asked to recall and draw the figures.
  Up to 2 points per figure. Scoring based on accuracy and placement of figure parts: A score of 0, 1 recognizable and incorrectly placed, 1 accurate or correctly placed or 2 both accurate and correctly placed; 0 is given if part is omitted or unrecognizable.
  Total possible 12 points
Benton Visual Memory Test; Trial 1 Immediate Recall 3 | Change from 1-Week to 1-Month after Series 1
  Immediate Recall for Visuospatial memory Min 0 and max 36; higher score better outcome Participant is presented with 6 figures. They are given 10 secs to view 6 pictures. Immediately asked to recall and draw the figures.
  Up to 2 points per figure. Scoring based on accuracy and placement of figure parts: A score of 0, 1 recognizable and incorrectly placed, 1 accurate or correctly placed or 2 both accurate and correctly placed; 0 is given if part is omitted or unrecognizable.
  Total possible 12 points
Benton Visual Memory Test; Trial 1 Immediate Recall 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Immediate Recall for Visuospatial memory Min 0 and max 36; higher score better outcome Participant is presented with 6 figures. They are given 10 secs to view 6 pictures. Immediately asked to recall and draw the figures.
  Up to 2 points per figure. Scoring based on accuracy and placement of figure parts: A score of 0, 1 recognizable and incorrectly placed, 1 accurate or correctly placed or 2 both accurate and correctly placed; 0 is given if part is omitted or unrecognizable.
  Total possible 12 points
Benton Visual Memory Test; Total Trials 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Total Trials 1-3. Learning Measure for Visuospatial memory Min 0 and max 36; higher score better outcome Total possible for each trial is 12 points. Sum of Total is learning score. Participant is presented with 6 figures. They are given 10 secs to view 6 pictures. Immediately asked to recall and draw the figures. This is repeated 3 times.
  Up to 2 points per figure. Scoring based on accuracy and placement of figure parts: A score of 0, 1 recognizable and incorrectly placed, 1 accurate or correctly placed or 2 both accurate and correctly placed; 0 is given if part is omitted or unrecognizable.
Benton Visual Memory Test; Total Trials 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Total Trials 1-3. Learning Measure for Visuospatial memory Min 0 and max 36; higher score better outcome Total possible for each trial is 12 points. Sum of Total is learning score. Participant is presented with 6 figures. They are given 10 secs to view 6 pictures. Immediately asked to recall and draw the figures. This is repeated 3 times.
  Up to 2 points per figure. Scoring based on accuracy and placement of figure parts: A score of 0, 1 recognizable and incorrectly placed, 1 accurate or correctly placed or 2 both accurate and correctly placed; 0 is given if part is omitted or unrecognizable.
Benton Visual Memory Test; Total Trials 3 | Change from 1-Week to 1-Month after Series 1
  Total Trials 1-3. Learning Measure for Visuospatial memory Min 0 and max 36; higher score better outcome Total possible for each trial is 12 points. Sum of Total is learning score. Participant is presented with 6 figures. They are given 10 secs to view 6 pictures. Immediately asked to recall and draw the figures. This is repeated 3 times.
  Up to 2 points per figure. Scoring based on accuracy and placement of figure parts: A score of 0, 1 recognizable and incorrectly placed, 1 accurate or correctly placed or 2 both accurate and correctly placed; 0 is given if part is omitted or unrecognizable.
Benton Visual Memory Test; Total Trials 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Total Trials 1-3. Learning Measure for Visuospatial memory Min 0 and max 36; higher score better outcome Total possible for each trial is 12 points. Sum of Total is learning score. Participant is presented with 6 figures. They are given 10 secs to view 6 pictures. Immediately asked to recall and draw the figures. This is repeated 3 times.
  Up to 2 points per figure. Scoring based on accuracy and placement of figure parts: A score of 0, 1 recognizable and incorrectly placed, 1 accurate or correctly placed or 2 both accurate and correctly placed; 0 is given if part is omitted or unrecognizable.
Benton Visual Memory Test; Delayed Recall 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Measures Delayed (20 minute) Recall for Visuospatial memory. {participant completes other tasks during delay) Min 0 and max 12; higher score better outcome Participant is asked to draw the figures from memory after a 20 minute delay (other tasks completed during this time).
  Total possible: 12 Scoring is based on accuracy and placement: 0 if unrecognizable or omitted, 1 recognizable, 1 either accurate or correctly placed or 2 both accurate and correctly placed, per figure.
Benton Visual Memory Test; Delayed Recall 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Measures Delayed (20 minute) Recall for Visuospatial memory. {participant completes other tasks during delay) Min 0 and max 12; higher score better outcome Participant is asked to draw the figures from memory after a 20 minute delay (other tasks completed during this time).
  Total possible: 12 Scoring is based on accuracy and placement: 0 if unrecognizable or omitted, 1 recognizable, 1 either accurate or correctly placed or 2 both accurate and correctly placed, per figure.
Benton Visual Memory Test; Delayed Recall 3 | Change from 1-Week to 1-Month after Series 1
  Measures Delayed (20 minute) Recall for Visuospatial memory. {participant completes other tasks during delay) Min 0 and max 12; higher score better outcome Participant is asked to draw the figures from memory after a 20 minute delay (other tasks completed during this time).
  Total possible: 12 Scoring is based on accuracy and placement: 0 if unrecognizable or omitted, 1 recognizable, 1 either accurate or correctly placed or 2 both accurate and correctly placed, per figure.
Benton Visual Memory Test; Delayed Recall 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Measures Delayed (20 minute) Recall for Visuospatial memory. {participant completes other tasks during delay) Min 0 and max 12; higher score better outcome Participant is asked to draw the figures from memory after a 20 minute delay (other tasks completed during this time).
  Total possible: 12 Scoring is based on accuracy and placement: 0 if unrecognizable or omitted, 1 recognizable, 1 either accurate or correctly placed or 2 both accurate and correctly placed, per figure.
Beck Depression Inventory (BDI) 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  21 item Questionnaire; Measures mood symptoms. Min 0 and max 63 0-13 minimal; 14-19 mild, 20-29 moderate, 30-63 severe; lower scores = better outcome Score per item: 1-3.
Beck Depression Inventory (BDI) 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  21 item Questionnaire; Measures mood symptoms. Min 0 and max 63 0-13 minimal; 14-19 mild, 20-29 moderate, 30-63 severe; lower scores = better outcome Score per item: 1-3.
Beck Depression Inventory (BDI) 3 | Change from 1-Week to 1-Month after Series 1
  21 item Questionnaire; Measures mood symptoms. Min 0 and max 63 0-13 minimal; 14-19 mild, 20-29 moderate, 30-63 severe; lower scores = better outcome Score per item: 1-3.
Beck Depression Inventory (BDI) 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  21 item Questionnaire; Measures mood symptoms. Min 0 and max 63 0-13 minimal; 14-19 mild, 20-29 moderate, 30-63 severe; lower scores = better outcome Score per item: 1-3.
Post Traumatic Stress Disorder (PCL) 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  17-item, symptom questionnaire Higher scores indicates greater endorsement of symptoms Min 17 and max 85 Reliable decrease 5-10 Clinically meaningful decrease 10-20 points Lower scores = better outcome Score ranges from 1-5 for each item.
Post Traumatic Stress Disorder (PCL) 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  17-item, symptom questionnaire Higher scores indicates greater endorsement of symptoms Min 17 and max 85 Reliable decrease 5-10 Clinically meaningful decrease 10-20 points Lower scores = better outcome Score ranges from 1-5 for each item.
Post Traumatic Stress Disorder (PCL) 3 | Change from 1-Week to 1-Month after Series 1
  17-item, symptom questionnaire Higher scores indicates greater endorsement of symptoms Min 17 and max 85 Reliable decrease 5-10 Clinically meaningful decrease 10-20 points Lower scores = better outcome Score ranges from 1-5 for each item.
Post Traumatic Stress Disorder (PCL) 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  17-item, symptom questionnaire Higher scores indicates greater endorsement of symptoms Min 17 and max 85 Reliable decrease 5-10 Clinically meaningful decrease 10-20 points Lower scores = better outcome Score ranges from 1-5 for each item.
Visual Analog Pain Rating Scale (VAS) 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Current Pain Rating scale of 1-10 Lower score = better outcome *must be lower than 7 at entry into study for study inclusion Participant rates current level of pain (includes body, muscular, headache etc) by marking a line on a continuous scale from 1-10.
Visual Analog Pain Rating Scale (VAS) 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Current Pain Rating scale of 1-10 Lower score = better outcome *must be lower than 7 at entry into study for study inclusion Participant rates current level of pain (includes body, muscular, headache etc) by marking a line on a continuous scale from 1-10.
Visual Analog Pain Rating Scale (VAS) 3 | Change from 1-Week to 1-Month after Series 1
  Current Pain Rating scale of 1-10 Lower score = better outcome *must be lower than 7 at entry into study for study inclusion Participant rates current level of pain (includes body, muscular, headache etc) by marking a line on a continuous scale from 1-10.
Visual Analog Pain Rating Scale (VAS) 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Current Pain Rating scale of 1-10 Lower score = better outcome *must be lower than 7 at entry into study for study inclusion Participant rates current level of pain (includes body, muscular, headache etc) by marking a line on a continuous scale from 1-10.
Short Form, McGill Pain Questionnaire 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Pain Rating (for the last 30 days) Min 0 and max 45; lower = better outcome Participant rates 15 categories of pain type (None = 0, mild = 1, moderate = 2, severe = 3).
  Sum totaled for all categories
Short Form, McGill Pain Questionnaire 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Pain Rating (for the last 30 days) Min 0 and max 45; lower = better outcome Participant rates 15 categories of pain type (None = 0, mild = 1, moderate = 2, severe = 3).
  Sum totaled for all categories
Short Form, McGill Pain Questionnaire 3 | Change from 1-Week to 1-Month after Series 1
  Pain Rating (for the last 30 days) Min 0 and max 45; lower = better outcome Participant rates 15 categories of pain type (None = 0, mild = 1, moderate = 2, severe = 3).
  Sum totaled for all categories
Short Form, McGill Pain Questionnaire 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Pain Rating (for the last 30 days) Min 0 and max 45; lower = better outcome Participant rates 15 categories of pain type (None = 0, mild = 1, moderate = 2, severe = 3).
  Sum totaled for all categories
Pittsburgh Sleep Quality Index (PSQI) 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  9 item questionnaire- made up of 7 component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction) Min of 0 and max of 3 per component. Global Sleep Score is total of 7 components Min score of 0 and max score of 21; lower score = better outcome
Pittsburgh Sleep Quality Index (PSQI) 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  9 item questionnaire- made up of 7 component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction) Min of 0 and max of 3 per component. Global Sleep Score is total of 7 components Min score of 0 and max score of 21; lower score = better outcome
Pittsburgh Sleep Quality Index (PSQI) 3 | Change from 1-Week to 1-Month after Series
  9 item questionnaire- made up of 7 component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction) Min of 0 and max of 3 per component. Global Sleep Score is total of 7 components Min score of 0 and max score of 21; lower score = better outcome
Pittsburgh Sleep Quality Index (PSQI) 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  9 item questionnaire- made up of 7 component scores (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction) Min of 0 and max of 3 per component. Global Sleep Score is total of 7 components Min score of 0 and max score of 21; lower score = better outcome
Quality of Community Integration Questionnaire Total CIQ Score 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  CIQ Cognitive Integration Score: 22 Questions Higher Score = better outcome Participant self-report of Current Level of Functional independence and satisfaction level of that ability on various cognitive and social/work/family interactions.
  Score 0-2 points for each item Composite Score: Sum of Home Integration 5 items, Social Integration 6 items and Productivity Scores 2 items; Range 0-29
Quality of Community Integration Questionnaire Total CIQ Score 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  CIQ Cognitive Integration Score: 22 Questions Higher Score = better outcome Participant self-report of Current Level of Functional independence and satisfaction level of that ability on various cognitive and social/work/family interactions.
  Score 0-2 points for each item Composite Score: Sum of Home Integration 5 items, Social Integration 6 items and Productivity Scores 2 items; Range 0-29
Quality of Community Integration Questionnaire Total CIQ Score 3 | Change from 1-Week to 1-Month after Series
  CIQ Cognitive Integration Score: 22 Questions Higher Score = better outcome Participant self-report of Current Level of Functional independence and satisfaction level of that ability on various cognitive and social/work/family interactions.
  Score 0-2 points for each item Composite Score: Sum of Home Integration 5 items, Social Integration 6 items and Productivity Scores 2 items; Range 0-29
Quality of Community Integration Questionnaire Total CIQ Score 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  CIQ Cognitive Integration Score: 22 Questions Higher Score = better outcome Participant self-report of Current Level of Functional independence and satisfaction level of that ability on various cognitive and social/work/family interactions.
  Score 0-2 points for each item Composite Score: Sum of Home Integration 5 items, Social Integration 6 items and Productivity Scores 2 items; Range 0-29
Quality of Community Integration Questionnaire (QCIQ) Score 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Quality of Community Integration (QCIQ) Score (Patient Satisfaction Level) 0-4 for satisfaction level on each item Range: 9 - 36 (Self-Report of satisfaction of home and social integration and productivity Higher Score = better outcome
Quality of Community Integration Questionnaire (QCIQ) Score 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Quality of Community Integration (QCIQ) Score (Patient Satisfaction Level) 0-4 for satisfaction level on each item Range: 9 - 36 (Self-Report of satisfaction of home and social integration and productivity Higher Score = better outcome
Quality of Community Integration Questionnaire (QCIQ) Score 3 | Change from 1-Week to 1-Month after Series
  Quality of Community Integration (QCIQ) Score (Patient Satisfaction Level) 0-4 for satisfaction level on each item Range: 9 - 36 (Self-Report of satisfaction of home and social integration and productivity Higher Score = better outcome
Quality of Community Integration Questionnaire (QCIQ) Score 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Quality of Community Integration (QCIQ) Score (Patient Satisfaction Level) 0-4 for satisfaction level on each item Range: 9 - 36 (Self-Report of satisfaction of home and social integration and productivity Higher Score = better outcome
Quality of Community Integration Questionnaire Cognitive Satisfaction Score 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Cognitive Satisfaction Score: Sum of 6 items related to cognitive satisfaction Range 6 - 24
Quality of Community Integration Questionnaire Cognitive Satisfaction Score 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Cognitive Satisfaction Score: Sum of 6 items related to cognitive satisfaction Range 6 - 24
Quality of Community Integration Questionnaire Cognitive Satisfaction Score 3 | Change from 1-Week to 1-Month after Series
  Cognitive Satisfaction Score: Sum of 6 items related to cognitive satisfaction Range 6 - 24
Quality of Community Integration Questionnaire Cognitive Satisfaction Score 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Cognitive Satisfaction Score: Sum of 6 items related to cognitive satisfaction Range 6 - 24
Quality of Community Integration Questionnaire Cognitive Quality of Life Score 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Cognitive Quality of Life Score:
  Cognitive Satisfaction Score x score on item 16. Range: 6 - 72
Quality of Community Integration Questionnaire Cognitive Quality of Life Score 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Cognitive Quality of Life Score:
  Cognitive Satisfaction Score x score on item 16. Range: 6 - 72
Quality of Community Integration Questionnaire Cognitive Quality of Life Score 3 | Change from 1-Week to 1-Month after Series
  Cognitive Quality of Life Score:
  Cognitive Satisfaction Score x score on item 16. Range: 6 - 72
Quality of Community Integration Questionnaire Cognitive Quality of Life Score 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Cognitive Quality of Life Score:
  Cognitive Satisfaction Score x score on item 16. Range: 6 - 72
Dysexecutive Functional Index (DEX) 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  Self-Report of psychosocial problems that participant may be experiencing in everyday life.
  20 Questions Scale of 0-4 for each item Total Possible: 80 Lower Score = better outcome
Dysexecutive Functional Index (DEX) 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  Self-Report of psychosocial problems that participant may be experiencing in everyday life.
  20 Questions Scale of 0-4 for each item Total Possible: 80 Lower Score = better outcome
Dysexecutive Functional Index (DEX) 3 | Change from 1-Week to 1-Month after Series
  Self-Report of psychosocial problems that participant may be experiencing in everyday life.
  20 Questions Scale of 0-4 for each item Total Possible: 80 Lower Score = better outcome
Dysexecutive Functional Index (DEX) 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  Self-Report of psychosocial problems that participant may be experiencing in everyday life.
  20 Questions Scale of 0-4 for each item Total Possible: 80 Lower Score = better outcome
Tinnitus Functional Index 1 | Change from Pre-Treatment Baseline to 1-Week after Series 1
  25 items; rated on a scale of 1-10 Lower score = better outcome Max = 10 per item; Max possible =250 overall Average across all valid responses Overall Score = Average*10 Max of 19 items must be marked >0 to be valid for tinnitus Subscores (each 3-4 items totaled) address 8 domains related to negative impact of tinnitus Intrusive, Sense of Control, Cognitive, Sleep, Auditory Difficulties, Relaxation, Quality of Life, and Emotional Distress
Tinnitus Functional Index 2 | Change from Pre-Treatment Baseline to 1-Month after Series 1
  25 items; rated on a scale of 1-10 Lower score = better outcome Max = 10 per item; Max possible =250 overall Average across all valid responses Overall Score = Average*10 Max of 19 items must be marked >0 to be valid for tinnitus Subscores (each 3-4 items totaled) address 8 domains related to negative impact of tinnitus Intrusive, Sense of Control, Cognitive, Sleep, Auditory Difficulties, Relaxation, Quality of Life, and Emotional Distress
Tinnitus Functional Index 3 | Change from 1-Week to 1-Month after Series
  25 items; rated on a scale of 1-10 Lower score = better outcome Max = 10 per item; Max possible =250 overall Average across all valid responses Overall Score = Average*10 Max of 19 items must be marked >0 to be valid for tinnitus Subscores (each 3-4 items totaled) address 8 domains related to negative impact of tinnitus Intrusive, Sense of Control, Cognitive, Sleep, Auditory Difficulties, Relaxation, Quality of Life, and Emotional Distress
Tinnitus Functional Index 4 | Change from Pre-Treatment Baseline to 1-Week after Series 2
  25 items; rated on a scale of 1-10 Lower score = better outcome Max = 10 per item; Max possible =250 overall Average across all valid responses Overall Score = Average*10 Max of 19 items must be marked >0 to be valid for tinnitus Subscores (each 3-4 items totaled) address 8 domains related to negative impact of tinnitus Intrusive, Sense of Control, Cognitive, Sleep, Auditory Difficulties, Relaxation, Quality of Life, and Emotional Distress

CONTACTS AND LOCATIONS:
Overall Officials: Paula I Martin, PhD, Principal Investigator — VA Boston Healthcare System, Jamaica Plain Campus, Boston, Ma
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
De-Identified data may be shared with written request and permission from VA Boston Healthcare System Internal Review Board, and Privacy Official.